CLINICAL TRIAL: NCT03567616
Title: A Phase 2, Open-Label, Multicenter, Dose-Escalation and Expansion Study of Venetoclax in Combination With Pomalidomide and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Venetoclax in Combination With Pomalidomide and Dexamethasone in Participants With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following results of the primary progression-free survival analysis from Study NCT02755597, company-sponsored MM studies were placed on partial clinical hold (PCH). Sponsor did not pursue release of the PCH for this study.
Sponsor: AbbVie (Industry)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-085; 2017-004232-11 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-06-12; First posted 2018-06-26 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Multiple Myeloma
Keywords: Cancer; Multiple Myeloma (MM); Relapsed or Refractory (R/R); Venetoclax; Pomalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Recurrence | interventions — venetoclax; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Dose Escalation (Experimental): Venetoclax (400 mg oral [PO], once daily [QD]) administered with pomalidomide (4 mg PO, QD) and dexamethasone (40 mg once weekly [qw]) in 28-day cycles until documented disease progression, documented unacceptable toxicity, withdrawal of consent, or the participant met other criteria for discontinuation per study protocol
  Interventions: Drug: Venetoclax; Drug: Pomalidomide; Drug: Dexamethasone
- Part 2: Dose Expansion, t(11;14) positive (Experimental): Participants positive for t(11;14) translocation were to receive the venetoclax dose determined to be safe in Part 1 as well as pomalidomide (4 mg oral [PO], once daily [QD]) and dexamethasone (40 mg once weekly [qw])
  Interventions: Drug: Venetoclax; Drug: Pomalidomide; Drug: Dexamethasone
- Part 2: Dose Expansion, t(11;14) negative (Experimental): Participants negative for t(11;14) translocation were to receive the venetoclax dose determined to be safe in Part 1 as well as pomalidomide (4 mg oral [PO], once daily [QD]) and dexamethasone (40 mg once weekly [qw])
  Interventions: Drug: Venetoclax; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Venetoclax — Tablet; oral
  Other Names: ABT-199; GDC-0199; Venclexta
Drug: Pomalidomide — Capsule; oral
  Other Names: Pomalyst
Drug: Dexamethasone — Administered orally; for participants over 75 years of age, dexamethasone could have been administered at a 20 mg dose [qw]

SUMMARY:
This was an open-label, multicenter study designed to evaluate the safety and preliminary efficacy of venetoclax combined with pomalidomide and dexamethasone in participants with relapsed or refractory (R/R) multiple myeloma (MM) who received at least 1 prior line of therapy with documented evidence of progression during or after the participant's last treatment regimen. The study was designed to consist of 2 parts: Part 1 (dose escalation) and Part 2 (dose expansion). For Part 2 the participants were to be divided into 2 cohorts, participants positive for t(11;14) translocation and participants negative for t(11;14) translocation.

DETAILED DESCRIPTION:
Following communication of the results of the primary progression-free survival (PFS) analysis from the Phase 3 BELLINI study (Study M14-031; NCT02755597), the company-sponsored MM studies were placed on partial clinical hold (PCH) in March 2019 by the United States (US) Food and Drug Administration and enrollment was halted. The sponsor did not pursue release of the PCH for this study; therefore, enrollment was not re-opened. In accordance with the terms of the PCH, participants who were deriving clinical benefit were allowed to continue to receive treatment. One participant was still active in Part 1 of the study when the sponsor decided not to pursue release of the PCH (in January 2020) and, therefore, continued to receive treatment and have regular assessments until disease progression. The study was discontinued when the last participant completed study treatment. No participants were enrolled in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory (R/R) multiple myeloma (MM) with documented evidence of progression during or after the participant's last treatment regimen
* Measurable disease as described in the protocol
* Received at least 1 prior line of therapy as described in the protocol
* Must meet prior antimyeloma treatment parameters, as described in the protocol, and includes:
* Received at least 2 consecutive cycles of lenalidomide or a lenalidomide-containing regimen
* Refractory to lenalidomide
* Exposed to a proteasome inhibitor (PI) alone or in combination with another agent
* Had a response of partial response (PR) or better to prior therapy based on the investigator's determination of response as defined by International Myeloma Working Group (IMWG) criteria
* Has t(11;14) status as described in the protocol and meets the following criteria:
* For Part 1: MM participants independent of cytogenetic profile
* For Part 2, Arm A: participant must be t(11;14) positive
* For Part 2, Arm B: participant must be t(11;14) negative
* An Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate kidney, liver and hematologic laboratory values

Exclusion Criteria:

* Previous treatment with venetoclax or other BCL-2 inhibitors, or previous treatment with pomalidomide
* Known sensitivity to any IMiDs
* Allogenic or syngeneic stem cell transplant within 6 months before the first dose of study drug or active ongoing graft versus host disease
* Autologous stem cell transplant within 12 weeks before the first dose of study drug
* Known meningeal involvement of MM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (11):
- United States (5):
  - John B. Amos Cancer Center - C /ID# 202055, Columbus, Georgia
  - University of Kansas Cancer Center /ID# 201292, Fairway, Kansas
  - Washington University-School of Medicine /ID# 201287, St Louis, Missouri
  - Duke University Hospital /ID# 200805, Durham, North Carolina
  - Ohio State Cancer Center /ID# 202443, Columbus, Ohio
- Spain (3):
  - Hospital Universitario Germans Trias i Pujol /ID# 200959, Badalona, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 200967, Barcelona
  - Hospital Clinico Universitario de Salamanca /ID# 200958, Salamanca
- United Kingdom (3):
  - Leicester Royal Infirmary /ID# 202238, Leicester, England
  - Norfolk and Norwich Univ Hosp /ID# 202240, Norwich, Norfolk
  - Univ Hospitals Birmingham NHS Foundation trust /ID# 203188, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Gasparetto C, Bowles KM, Abdallah AO, Morris L, Mander G, Coppola S, Wang J, Ross JA, Bueno OF, Arriola E, Mateos MV. A Phase II Study of Venetoclax in Combination With Pomalidomide and Dexamethasone in Relapsed/Refractory Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2021 Nov;21(11):775-784. doi: 10.1016/j.clml.2021.07.029. Epub 2021 Aug 1. PMID 34551886
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set: participants who received at least 1 dose of study drug
Groups:
- All Participants: Participants who received at least 1 dose of study drug (venetoclax 400 mg, pomalidomide 4 mg, and dexamethasone 40 mg)
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 0
Not Completed | 8
Not completed — Disease progression | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who received at least 1 dose of study drug
Groups:
- Participants Positive for t(11;14) Translocation: Participants positive for t(11;14) translocation who received at least 1 dose of study drug (venetoclax 400 mg, pomalidomide 4 mg, and dexamethasone 40 mg)
- Participants Negative for t(11;14) Translocation: Participants negative for t(11;14) translocation who received at least 1 dose of study drug (venetoclax 400 mg, pomalidomide 4 mg, and dexamethasone 40 mg)
- Total: Total of all reporting groups
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 68.0 [67 to 74] | 66.0 [60 to 77] | 67.5 [60 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 7
  Black/African American | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to 70 weeks)
Population: Safety Analysis Set: participants who received at least 1 dose of study drug (venetoclax 400 mg, pomalidomide 4 mg, and dexamethasone 40 mg)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation
Number analyzed (Participants) | 3 | 5
Participants
  Any TEAE | 3 | 5
  TESAE | 3 | 2

2. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants experiencing a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) using the International Myeloma Working Group (IMWG) 2016 criteria for disease response and progression. CR= negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow; sCR= CR + normal serum free light chain (FLC) ratio and absence of clonal cells in bone marrow; VGPR= serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein level + urine M-protein level < 100 mg per 24 hours; PR= ≥ 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours.
Time Frame: Approximately 15 months
Population: Full Analysis Set: participants who received at least 1 dose of study drug (venetoclax 400 mg, pomalidomide 4 mg, and dexamethasone 40 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation | All Participants
Number analyzed (Participants) | 3 | 5 | 8
percentage of participants | 66.7 [9.4 to 99.2] | 60.0 [14.7 to 94.7] | 62.5 [24.5 to 91.5]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the number of days from the date of first dose of any study drug to the date of disease progression or death, whichever occurs first. All disease progression was to be included regardless of whether the event occurred during or after the participant was taking any study drug.
Time Frame: Approximately 20 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation | All Participants
Number analyzed (Participants) | 3 | 5 | 8
days | 220.0 [11.0 to NA] — Not calculable/estimable due to low number of participants with events | NA [57.0 to NA] — Not calculable/estimable due to low number of participants with events | 320.0 [11.0 to NA] — Not calculable/estimable due to low number of participants with events

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR for a given participant is defined as the number of days from the date of that participant's first documented response (Partial Response [PR] or better) to the date of first documented disease progression (PD) or death due to multiple myeloma (MM), whichever occurs first. If the participant with a documented response did not have an event of PD and the participant had not died due to MM, the participant's data was to be censored.
Time Frame: Approximately 15 months
Population: Full Analysis Set: participants who received at least 1 dose of study drug (venetoclax 400 mg, pomalidomide 4 mg, and dexamethasone 40 mg) and had disease progression or death due to multiple myeloma
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation | All Participants
Number analyzed (Participants) | 2 | 3 | 5
days | 393.0 [NA to NA] — Not calculable/estimable due to low number of participants with events | NA [NA to NA] — Not calculable/estimable due to low number of participants with events | 393.0 [NA to NA] — Not calculable/estimable due to low number of participants with events

5. Secondary Outcome: Time-to-progression (TTP)
Description: TTP for a given participant is defined as the number of days from the date of first dose to the date of first documented disease progression (PD) or death due to multiple myeloma (MM), whichever occurs first. If the participant did not have an event of PD and the participant had not died due to MM, the participant's data was to be censored.
Time Frame: Approximately 15 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation | All Participants
Number analyzed (Participants) | 3 | 5 | 8
days | 420.0 [NA to NA] — Not calculable/estimable due to low number of participants with events | NA [57.0 to NA] — Not calculable/estimable due to low number of participants with events | 420.0 [57.0 to NA] — Not calculable/estimable due to low number of participants with events

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after last study drug administration, up to 70 weeks.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 30 days have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Participants Positive for t(11;14) Translocation | Participants Negative for t(11;14) Translocation
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Positive for t(11;14) Translocation (N=3) | Participants Negative for t(11;14) Translocation (N=5)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
PNEUMOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 0 (0)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Positive for t(11;14) Translocation (N=3) | Participants Negative for t(11;14) Translocation (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (3) | 2 (14)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (6)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (10) | 4 (34)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (6)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (2)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (2)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 2 (3) | 2 (3)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (2)
PYREXIA (General disorders) | 1 (1) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (2)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (3)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 2 (2)
BLOOD IMMUNOGLOBULIN G DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 2 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 1 (5)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (2)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 2 (15)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 1 (2)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 1 (1)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (2) | 1 (2)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03567616/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03567616/SAP_001.pdf